CLINICAL TRIAL: NCT06119906
Title: Prospective Pilot Cohort Study to Assess Early Diagnostic Utility of Hyper-Spectral Endoscopy for Detection of Neoplasia in Barrett's Oesophagus
Brief Title: Hyper-Spectral Endoscopy for Detection of Early Neoplasia in Barrett's Oesophagus
Acronym: HySE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Cambridge (Other)
Collaborators: University of Manchester (Other)
Responsible Party: Principal Investigator, Massimiliano di Pietro, MD, Principal Investigator, University of Cambridge
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HySe trial v1.0
Record Dates: First submitted 2023-10-16; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Standard + Experimental Endoscopy (Experimental): The endoscopist will intubate the patient with a high resolution white light endoscope (Olympus GIFH290Z or GIF-EZ1500) and thoroughly inspect the mucosal surface of the oesophagus. A careful note will be made of any visible lesion with their location, and the surrounding mucosa will be marked with cautery to localize the lesion for further hyperspectral imaging and biopsy. We will aim to identify at least two areas of interest per patient with the possibility to select more if the length of the Barrett's oesophagus allows. The endoscopist will remove the standard of care endoscope and then reintubate the patient with the experimental device and perform unbiased imaging first followed by targeted imaging of the endoscopic areas previously marked
  Interventions: Device: Hyper-Spectral Endoscopy

INTERVENTIONS:
Device: Hyper-Spectral Endoscopy — We have developed a custom hyperspectral endoscopy approach based around a commercially available endoscopy system. An Olympus gastroscope (GIF-H260) and video processor and display are used with a modified light source that incorporates a laser with tunable wavelength for illuminating the scene through the endoscope. A live video feed from the gastroscope is displayed on the endoscopy monitors and can be acquired and saved in the native video acquisition system. The spectral imaging data is also saved within this video feed, where imaging wavelength corresponds to a given timestamp in the video.

SUMMARY:
The goal of this clinical trial is to assess the efficacy of hyperspectral endoscopic imaging to distinguish neoplasia from non-dysplastic Barrett's oesophagus in vivo. The main outcome measures are: 1) Classification of spectral patterns corresponding to neoplastic vs non-neoplastic Barrett's; 2) Image quality assessed by the endoscopist by VAS rating the level of confidence in delineating the area of interest; 3) Time to perform hyperspectral imaging; 4) Quantification of molecular biomarkers in endoscopic areas with neoplastic spectral patterns.

Participants will firstly undergo a standard endoscopy, followed by another endoscopy using the experimental HySe device. Subsequently, patients will receive biopsies according to Seattle protocol, and up to 6 additional (optional) snap frozen research biopsies.

DETAILED DESCRIPTION:
This trial is designed to evaluate the feasibility of hyperspectral endoscopic imaging in vivo.

The team has developed a custom hyperspectral endoscope based around a commercially available, standard-of-care endoscopy stack from Olympus (Tokyo, Japan). In this system, the original gastroscope, video processor and display are used with a modified light source that incorporates a laser with tunable wavelength for illuminating the scene through the endoscope. A live video feed from the gastroscope is displayed on the endoscopy theatre monitors and can be acquired and saved in the native video acquisition system.

Given that it is essential in the pilot study to assess the detection of neoplastic lesions in a small patient cohort, we will artificially enrich for patients with early neoplasia by including patients with previously recognized early neoplasia within Barrett's oesophagus (high grade dysplasia and intramucosal adenocarcinoma). These patients will receive a clinically indicated endoscopy to be assessed to determine eligibility for endoscopic treatment, and imaging would be done at this time point. This will allow the team to have sufficient number of outcomes to have preliminary data on diagnostic accuracy and be able to power future studies in non-enriched patient cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects over 18 years.
* Previous diagnosis of Barrett's oesophagus, with an endoscopic length of at least 2 cm if circumferential (C≥2 according to Prague classification) or 3 cm if not circumferential (maximal extent M≥3, according to Prague classification).
* Previous diagnosis of oesophageal glandular dysplasia or early oesophageal adenocarcinoma for consideration of endoscopic therapy.

Exclusion Criteria:

* History of oesophageal stricture precluding passage of the endoscope.
* Pregnancy, or planned pregnancy during the course of the study.
* Currently breastfeeding.
* Any history of oesophageal varices, liver impairment of moderate or worse severity (Child's- Pugh class B & C) or evidence of varices on initial treatment endoscopy.
* Any history of oesophageal surgery, except for uncomplicated fundoplication.
* History of coagulopathy, with INR>1.3 and/or platelet count of <75,000.
* On clopidogrel, and/or warfarin for high risk condition and unable to withhold temporarily the medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Contrast of neoplastic vs non-neoplastic Barrett's | Post-hoc analysis after the endoscopy - time scale 6-12 months from procedure
  Pixel intensity value at 16 different wave lengths in endoscopic areas of interest as compared with standard-of-care RGB white light endoscopy

SECONDARY OUTCOMES:
Image quality of Hyper-Spectral Endoscopy in vivo | Immediately after the intervention
  Visual analogue scale (VAS) rating the level of confidence in delineating the area of interest
Time to perform hyperspectral imaging | During the intervention
  Time in Minutes
Quantification of molecular biomarkers in endoscopic areas with neoplastic spectral patterns | Post-hoc analysis after the endoscopy - time scale 6-12 months from procedure
  Intensity of staining of Immunohistochemical markers
Image quality of Hyper-Spectral Endoscopy after post-hoc analysis | Post-hoc analysis after the endoscopy - time scale 6-12 months from procedure
  Visual analogue scale (VAS) rating the level of confidence in delineating the area of interest

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Bohndiek, Principal Investigator — University of Cambridge
Locations (1):
- Cambridge University Hospital, Cambridge, County (optional), United Kingdom

IPD SHARING:
Plan to Share IPD: No